CLINICAL TRIAL: NCT02117934
Title: A Phase 3, Observer-Blinded, Randomized, Active-Controlled (Engerix-B), Multicenter Trial of the Safety and Immunogenicity of HEPLISAV in Adults 18 to 70 Years of Age
Brief Title: Safety and Immunogenicity Study of the Hepatitis B Vaccine, HEPLISAV™, Compared to Engerix-B® Vaccine
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Dynavax Technologies Corporation (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Prevention
Other Study IDs: DV2-HBV-23
Record Dates: First submitted 2014-04-15; First posted 2014-04-21 (Estimated); Results first posted 2018-01-10 (Actual); Last update posted 2019-03-20 (Actual); Status verified 2019-03

CONDITIONS: Healthy
Keywords: HBV vaccine; HEPLISAV-B; Hepatitis B vaccine; Hepatitis B; Hepatitis; Hepatitis B virus (HBV); Prevention and Control; Healthy; Healthy volunteers
MeSH Terms: conditions — Hepatitis B; Hepatitis | interventions — Hepatitis B Vaccines; Heplisav-B; Engerix-B

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (2):
- HEPLISAV (Experimental): 0.5 mL HEPLISAV (20 mcg HBsAg and 3000 mcg 1018) administered intramuscularly in the deltoid muscle at Weeks 0, 4, and placebo (saline injection) at Week 24, followed by a 52-week safety follow-up from the last active dose of HEPLISAV.
  Interventions: Biological: HEPLISAV
- Engerix-B (Active Comparator): 1.0 mL Engerix-B (20 mcg HBsAg adsorbed on 500 mcg of aluminum hydroxide) administered intramuscularly in the deltoid muscle at Weeks 0, 4, and 24, followed by a 32-week safety follow-up from the last dose of Engerix-B.
  Interventions: Biological: Engerix-B

INTERVENTIONS:
Biological: HEPLISAV — Intramuscular injections at Week 0 and Week 4, plus a placebo injection at Week 24
  Other Names: Hepatitis B vaccine (recombinant), adjuvanted; HEPLISAV-B
  Arms: HEPLISAV
Biological: Engerix-B — Intramuscular injections at Week 0, Week 4, and Week 24
  Other Names: Hepatitis B vaccine (recombinant)
  Arms: Engerix-B

SUMMARY:
The purpose of the study is to evaluate the safety and immunogenicity of an investigational hepatitis B vaccine (HEPLISAV) in adults 18 to 70 years of age.

ELIGIBILITY:
A subject must meet all of the following criteria to be eligible for the trial:

Inclusion Criteria:

* Be 18-70 years of age, inclusive
* Able to comprehend and follow all required study procedures and be available for all visits scheduled in the study
* If a woman is of childbearing potential, she must consistently use an acceptable method of contraception or confirm in writing she will abstain from sexual activity from the Screening Visit through Week 28.
* Able and willing to provide informed consent

A subject with any one of the following criteria is not eligible for the trial:

Exclusion Criteria:

* Previous receipt of any hepatitis B vaccine
* History of hepatitis B or human immunodeficiency virus (HIV) infection or positive test for HBsAg, anti-HBs, antibody to hepatitis B core antigen (anti-HBc), or antibody to HIV
* History of autoimmune disorder
* History of sensitivity to any component of study vaccines
* Has received the following prior to the first injection:

  1. Within 28 days:

     * Any vaccine
     * Systemic corticosteroids (more than 3 consecutive days) or other immunomodulators or immune suppressive medication
     * Granulocyte colony-stimulating factor (G-CSF) or granulocyte-macrophage colony-stimulating factor (GM-CSF)
     * Any other investigational medicinal agent
  2. Within 90 days: Blood products or immunoglobulin
  3. At any time: An injection of DNA plasmids or oligonucleotide
* If female: Pregnant, nursing, or planning to become pregnant during the trial
* Is undergoing chemotherapy or expected to receive chemotherapy during the study period; has a diagnosis of cancer within the last 5 years other than squamous or basal cell carcinoma of the skin
* Any other medical condition considered by the investigator likely to interfere with the subject's compliance or the interpretation of study assessments

Ages: 18 Years to 70 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 8374 (Actual)
Dates: Start 2014-04; Primary Completion 2015-10 (Actual); Study Completion 2015-10 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Robert Janssen, MD, Study Director — Dynavax Technologies Corporation
Locations (37):
- United States (37):
  - Clinical Research Advantage, Inc., Birmingham, Alabama
  - Clinical Research Advantage, Inc., Chandler, Arizona
  - Radiant Research, Chandler, Arizona
  - Clinical Research Advantage, Inc., Glendale, Arizona
  - Clinical Research Advantage, Inc., Mesa, Arizona
  - Clinical Research Advantage, Inc., Phoenix, Arizona
  - Radiant Research, Scottsdale, Arizona
  - Clinical Research Advantage, Inc., Tempe, Arizona
  - Radiant Research, Tucson, Arizona
  - Clinical Research Advantage, Inc., Tucson, Arizona
  - Radiant Research, Santa Rosa, California
  - Clinical Research Advantage, Inc., Vista, California
  - Clinical Research Advantage, Inc., Centennial, Colorado
  - Clinical Research Advantage, Inc., Colorado Springs, Colorado
  - Radiant Research, Denver, Colorado
  - Radiant Research, Pinellas Park, Florida
  - Radiant Research, Atlanta, Georgia
  - Radiant Research, Chicago, Illinois
  - Clinical Research Advantage, Inc, Evansville, Indiana
  - Clinical Research Advantage, Inc., Council Bluffs, Iowa
  - Radiant Research, Edina, Minnesota
  - Radiant Research, St Louis, Missouri
  - Clinical Research Advantage, Inc., Elkhorn, Nebraska
  - Clinical Research Advantage, Inc., Fremont, Nebraska
  - Clinical Research Advantage, Inc., Omaha, Nebraska
  - Clinical Research Advantage, Inc., Henderson, Nevada
  - Clinical Research Advantage, Inc., Las Vegas, Nevada
  - Radiant Research, Akron, Ohio
  - Radiant Research, Cincinnati, Ohio
  - Radiant Research, Columbus, Ohio
  - Clinical Research Advantage, Inc., Anderson, South Carolina
  - Radiant Research, Anderson, South Carolina
  - Radiant Research, Greer, South Carolina
  - Radiant Research, Dallas, Texas
  - Clinical Research Advantage, Inc., Plano, Texas
  - Radiant Research, San Antonio, Texas
  - Radiant Research, Murray, Utah

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Hyer RN, Janssen RS. Immunogenicity and safety of a 2-dose hepatitis B vaccine, HBsAg/CpG 1018, in persons with diabetes mellitus aged 60-70 years. Vaccine. 2019 Sep 16;37(39):5854-5861. doi: 10.1016/j.vaccine.2019.08.005. Epub 2019 Aug 17. PMID 31431412
- [Derived] Jackson S, Lentino J, Kopp J, Murray L, Ellison W, Rhee M, Shockey G, Akella L, Erby K, Heyward WL, Janssen RS; HBV-23 Study Group. Immunogenicity of a two-dose investigational hepatitis B vaccine, HBsAg-1018, using a toll-like receptor 9 agonist adjuvant compared with a licensed hepatitis B vaccine in adults. Vaccine. 2018 Jan 29;36(5):668-674. doi: 10.1016/j.vaccine.2017.12.038. Epub 2017 Dec 27. PMID 29289383

RESULTS

PARTICIPANT FLOW:
Groups:
- HEPLISAV: 0.5 mL HEPLISAV (20 mcg HBsAg and 3000 mcg 1018)
  HEPLISAV and/or Placebo: Intramuscular (IM) injections at Week 0, Week 4, plus a placebo (saline) injection at Week 24
- Engerix-B: 1.0 mL Engerix-B
  Engerix-B: Intramuscular injections at Week 0, Week 4, and Week 24
Period: Overall Study
Arm/Group | HEPLISAV | Engerix-B
Started | 5592 | 2782
Completed | 5092 | 2567
Not Completed | 500 | 215

BASELINE CHARACTERISTICS:
Population: Safety Population: All subjects who received at least 1 study injection and who had any post-baseline safety data
Groups:
- Total: Total of all reporting groups
Arm/Group | HEPLISAV | Engerix-B | Total
Number analyzed (Participants) | 5587 | 2781 | 8368
Age, Customized [Count of Participants; unit: Participants]
  Age ≥ 18 to ≤ 39 years | 1132 | 561 | 1693
  Age ≥ 40 years | 4455 | 2220 | 6675
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 2743 | 1390 | 4133
  Male | 2844 | 1391 | 4235
Region of Enrollment [Count of Participants; unit: Participants]
  United States | 5587 | 2781 | 8368

OUTCOME MEASURES:

1. Primary Outcome: Percentage of Subjects Reporting Clinically Significant Adverse Events - Medically-attended Adverse Events, Serious Adverse Events, and Immune-mediated Adverse Events of Special Interest
Description: The percentage of participants with Medically-attended adverse events (MAEs), Serious Adverse Events (SAEs), and immune-mediated Adverse Events of Special Interest (AESIs). MAEs are Adverse events (AEs) for which a subject sought medical attention at a doctor's office, clinic or study site, or emergency room, or was hospitalized. SAEs are AEs that met the definition of Serious per FDA regulations. Immune-mediated AESIs are AEs that were confirmed to be autoimmune in etiology.
Time Frame: Week 56
Population: Safety Population: All participants who received at least 1 study injection and who had any post-baseline safety data
Measure: Number; unit: percentage of participants
Arm/Group | HEPLISAV | Engerix-B
Number analyzed (Participants) | 5587 | 2781
percentage of participants
  New-onset Immune-mediated Adverse Events | 0.1 | 0.04
  Medically-attended Adverse Events | 46.0 | 46.2
  Serious Adverse Events | 6.2 | 5.3

2. Primary Outcome: Percentage of Subjects With Type 2 Diabetes Mellitus Who Have a Seroprotective Immune Response
Description: Percentage of subjects with type 2 diabetes mellitus who have a seroprotective immune response (anti-HBs ≥ 10 milli-international unit (mIU)/mL) who receive HEPLISAV compared with subjects who receive Engerix-B
Time Frame: Week 28
Population: Per-Protocol Diabetes Population:Randomized subjects with type 2 diabetes mellitus (clinical diagnosis of T2DM taking at least oral or non-insulin injectable hypoglycemic agent and/or insulin) who received all study injections, had no major protocol deviations, and had anti-HBs levels obtained within the study visit window at Week 28.
Measure: Number (95% Confidence Interval); unit: Percentage of participants
Arm/Group | HEPLISAV | Engerix-B
Number analyzed (Participants) | 640 | 321
Percentage of participants | 90.0 [87.4 to 92.2] | 65.1 [59.6 to 70.3]

ADVERSE EVENTS:
Time Frame: Through Week 56
Description: Adverse Events were assessed for the Safety Population: All participants who received at least 1 study injection and who had any post-baseline safety data.
Arm/Group | HEPLISAV | Engerix-B
Serious Adverse Events (participants affected / at risk) | 345/5587 | 148/2781
Other Adverse Events (participants affected / at risk) | 1097/5587 | 549/2781
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | HEPLISAV (N=5587) | Engerix-B (N=2781)
Anaemia (Blood and lymphatic system disorders) | 2 | 1
Anaemia vitamin b12 deficiency (Blood and lymphatic system disorders) | 0 | 1
Leukocytosis (Blood and lymphatic system disorders) | 1 | 0
Microcytic anaemia (Blood and lymphatic system disorders) | 1 | 0
Acute coronary syndrome (Cardiac disorders) | 1 | 0
Acute myocardial infarction (Cardiac disorders) | 14 | 1
Angina pectoris (Cardiac disorders) | 2 | 1
Angina unstable (Cardiac disorders) | 1 | 0
Atrial fibrillation (Cardiac disorders) | 6 | 3
Atrial flutter (Cardiac disorders) | 2 | 1
Bradycardia (Cardiac disorders) | 2 | 0
Cardiac arrest (Cardiac disorders) | 3 | 0
Cardiac failure (Cardiac disorders) | 2 | 0
Cardiac failure acute (Cardiac disorders) | 1 | 0
Cardiac failure congestive (Cardiac disorders) | 6 | 3
Cardiac ventricular thrombosis (Cardiac disorders) | 1 | 1
Cardio-respiratory arrest (Cardiac disorders) | 1 | 1
Cardiogenic shock (Cardiac disorders) | 1 | 0
Cardiomyopathy (Cardiac disorders) | 0 | 1
Coronary artery disease (Cardiac disorders) | 6 | 2
Coronary artery occlusion (Cardiac disorders) | 1 | 1
Coronary artery stenosis (Cardiac disorders) | 2 | 0
Hypertensive heart disease (Cardiac disorders) | 4 | 1
Myocardial infarction (Cardiac disorders) | 2 | 1
Myocardial ischaemia (Cardiac disorders) | 1 | 0
Pulseless electrical activity (Cardiac disorders) | 1 | 0
Supraventricular tachycardia (Cardiac disorders) | 1 | 0
Ventricular fibrillation (Cardiac disorders) | 1 | 0
Ventricular tachycardia (Cardiac disorders) | 2 | 0
Atrial septal defect (Congenital, familial and genetic disorders) | 1 | 0
Ebstein's anomaly (Congenital, familial and genetic disorders) | 1 | 1
Sickle cell anaemia with crisis (Congenital, familial and genetic disorders) | 1 | 0
Vertigo (Ear and labyrinth disorders) | 1 | 0
Vertigo positional (Ear and labyrinth disorders) | 1 | 1
Inappropriate antidiuretic hormone secretion (Endocrine disorders) | 1 | 0
Pituitary-dependent cushing's syndrome (Endocrine disorders) | 0 | 1
Thyroid mass (Endocrine disorders) | 0 | 1
Abdominal hernia (Gastrointestinal disorders) | 1 | 0
Abdominal pain (Gastrointestinal disorders) | 2 | 2
Appendix disorder (Gastrointestinal disorders) | 1 | 0
Colitis (Gastrointestinal disorders) | 2 | 0
Colitis ulcerative (Gastrointestinal disorders) | 1 | 0
Constipation (Gastrointestinal disorders) | 2 | 1
Cyclic vomiting syndrome (Gastrointestinal disorders) | 1 | 0
Diarrhoea (Gastrointestinal disorders) | 1 | 0
Diverticular perforation (Gastrointestinal disorders) | 2 | 1
Diverticulum intestinal haemorrhagic (Gastrointestinal disorders) | 1 | 0
Duodenal ulcer haemorrhage (Gastrointestinal disorders) | 0 | 1
Gastric ulcer (Gastrointestinal disorders) | 0 | 1
Gastric ulcer haemorrhage (Gastrointestinal disorders) | 1 | 0
Gastritis (Gastrointestinal disorders) | 2 | 0
Gastritis alcoholic (Gastrointestinal disorders) | 1 | 0
Gastritis alcoholic haemorrhagic (Gastrointestinal disorders) | 1 | 0
Gastritis haemorrhagic (Gastrointestinal disorders) | 1 | 0
Gastrointestinal haemorrhage (Gastrointestinal disorders) | 2 | 1
Gastrooesophageal reflux disease (Gastrointestinal disorders) | 3 | 1
Ileus (Gastrointestinal disorders) | 1 | 0
Ileus paralytic (Gastrointestinal disorders) | 1 | 0
Impaired gastric emptying (Gastrointestinal disorders) | 0 | 1
Inguinal hernia (Gastrointestinal disorders) | 0 | 1
Intestinal obstruction (Gastrointestinal disorders) | 0 | 1
Large intestine perforation (Gastrointestinal disorders) | 1 | 1
Lower gastrointestinal haemorrhage (Gastrointestinal disorders) | 0 | 1
Oesophageal spasm (Gastrointestinal disorders) | 1 | 0
Oesophagitis (Gastrointestinal disorders) | 1 | 0
Pancreatitis (Gastrointestinal disorders) | 2 | 0
Pancreatitis acute (Gastrointestinal disorders) | 1 | 2
Rectal haemorrhage (Gastrointestinal disorders) | 1 | 2
Rectal prolapse (Gastrointestinal disorders) | 1 | 0
Small intestinal obstruction (Gastrointestinal disorders) | 6 | 2
Upper gastrointestinal haemorrhage (Gastrointestinal disorders) | 2 | 0
Varices oesophageal (Gastrointestinal disorders) | 1 | 0
Chest pain (General disorders) | 2 | 1
Death (General disorders) | 2 | 0
Device failure (General disorders) | 1 | 0
Drug withdrawal syndrome (General disorders) | 0 | 1
Non-cardiac chest pain (General disorders) | 9 | 7
Bile duct stone (Hepatobiliary disorders) | 2 | 1
Cholecystitis (Hepatobiliary disorders) | 5 | 2
Cholecystitis acute (Hepatobiliary disorders) | 0 | 2
Cholecystitis chronic (Hepatobiliary disorders) | 1 | 2
Cholelithiasis (Hepatobiliary disorders) | 4 | 4
Hepatic cirrhosis (Hepatobiliary disorders) | 1 | 1
Ischaemic hepatitis (Hepatobiliary disorders) | 1 | 0
Hypersensitivity (Immune system disorders) | 1 | 1
Abscess limb (Infections and infestations) | 1 | 0
Abscess neck (Infections and infestations) | 1 | 0
Appendicitis (Infections and infestations) | 3 | 1
Appendicitis perforated (Infections and infestations) | 2 | 0
Arthritis bacterial (Infections and infestations) | 1 | 0
Bacteraemia (Infections and infestations) | 1 | 0
Bronchitis (Infections and infestations) | 3 | 0
Cellulitis (Infections and infestations) | 7 | 4
Cellulitis of male external genital organ (Infections and infestations) | 1 | 0
Cellulitis orbital (Infections and infestations) | 0 | 1
Cholecystitis infective (Infections and infestations) | 1 | 0
Clostridium difficile colitis (Infections and infestations) | 1 | 0
Device related infection (Infections and infestations) | 1 | 0
Diabetic foot infection (Infections and infestations) | 2 | 1
Diverticulitis (Infections and infestations) | 1 | 2
Erysipelas (Infections and infestations) | 0 | 1
Gastroenteritis (Infections and infestations) | 4 | 1
Gastroenteritis viral (Infections and infestations) | 0 | 1
Groin abscess (Infections and infestations) | 1 | 1
Hepatitis c (Infections and infestations) | 2 | 0
Infectious colitis (Infections and infestations) | 2 | 0
Influenza (Infections and infestations) | 2 | 1
Latent tuberculosis (Infections and infestations) | 1 | 0
Lobar pneumonia (Infections and infestations) | 2 | 0
Meningitis (Infections and infestations) | 2 | 0
Mycobacterium avium complex infection (Infections and infestations) | 1 | 0
Osteomyelitis (Infections and infestations) | 1 | 1
Otitis media bacterial (Infections and infestations) | 1 | 0
Periorbital cellulitis (Infections and infestations) | 1 | 0
Perirectal abscess (Infections and infestations) | 1 | 1
Pneumonia (Infections and infestations) | 15 | 8
Pneumonia escherichia (Infections and infestations) | 1 | 0
Pneumonia staphylococcal (Infections and infestations) | 1 | 0
Post procedural infection (Infections and infestations) | 0 | 1
Postoperative wound infection (Infections and infestations) | 0 | 1
Pyelonephritis (Infections and infestations) | 2 | 1
Pyelonephritis acute (Infections and infestations) | 2 | 0
Sepsis (Infections and infestations) | 5 | 1
Splenic abscess (Infections and infestations) | 1 | 0
Staphylococcal abscess (Infections and infestations) | 1 | 1
Staphylococcal osteomyelitis (Infections and infestations) | 0 | 1
Upper respiratory tract infection (Infections and infestations) | 1 | 0
Urinary tract infection (Infections and infestations) | 0 | 1
Urinary tract infection enterococcal (Infections and infestations) | 1 | 0
Urosepsis (Infections and infestations) | 4 | 2
Viral sepsis (Infections and infestations) | 1 | 0
Wound infection (Infections and infestations) | 0 | 1
Wound infection staphylococcal (Infections and infestations) | 1 | 0
Accident (Injury, poisoning and procedural complications) | 1 | 0
Accidental overdose (Injury, poisoning and procedural complications) | 1 | 0
Ankle fracture (Injury, poisoning and procedural complications) | 1 | 1
Arterial injury (Injury, poisoning and procedural complications) | 1 | 0
Cervical vertebral fracture (Injury, poisoning and procedural complications) | 1 | 1
Concussion (Injury, poisoning and procedural complications) | 1 | 0
Craniocerebral injury (Injury, poisoning and procedural complications) | 0 | 1
Facial bones fracture (Injury, poisoning and procedural complications) | 0 | 1
Femoral neck fracture (Injury, poisoning and procedural complications) | 0 | 2
Femur fracture (Injury, poisoning and procedural complications) | 2 | 0
Foot fracture (Injury, poisoning and procedural complications) | 1 | 0
Forearm fracture (Injury, poisoning and procedural complications) | 0 | 1
Gastrointestinal anastomotic leak (Injury, poisoning and procedural complications) | 0 | 1
Gun shot wound (Injury, poisoning and procedural complications) | 3 | 0
Hand fracture (Injury, poisoning and procedural complications) | 1 | 0
Head injury (Injury, poisoning and procedural complications) | 0 | 1
Hip fracture (Injury, poisoning and procedural complications) | 2 | 0
Humerus fracture (Injury, poisoning and procedural complications) | 2 | 0
Intentional overdose (Injury, poisoning and procedural complications) | 1 | 0
Jaw fracture (Injury, poisoning and procedural complications) | 1 | 0
Laceration (Injury, poisoning and procedural complications) | 1 | 1
Lower limb fracture (Injury, poisoning and procedural complications) | 1 | 0
Lumbar vertebral fracture (Injury, poisoning and procedural complications) | 2 | 0
Overdose (Injury, poisoning and procedural complications) | 1 | 0
Patella fracture (Injury, poisoning and procedural complications) | 2 | 0
Peripheral nerve injury (Injury, poisoning and procedural complications) | 1 | 0
Post procedural haematoma (Injury, poisoning and procedural complications) | 2 | 0
Postoperative fever (Injury, poisoning and procedural complications) | 1 | 1
Postoperative ileus (Injury, poisoning and procedural complications) | 1 | 1
Procedural intestinal perforation (Injury, poisoning and procedural complications) | 1 | 0
Procedural pain (Injury, poisoning and procedural complications) | 0 | 2
Rib fracture (Injury, poisoning and procedural complications) | 2 | 0
Scapula fracture (Injury, poisoning and procedural complications) | 1 | 0
Seroma (Injury, poisoning and procedural complications) | 1 | 0
Spinal fracture (Injury, poisoning and procedural complications) | 1 | 0
Stab wound (Injury, poisoning and procedural complications) | 1 | 0
Tibia fracture (Injury, poisoning and procedural complications) | 1 | 0
Toxicity to various agents (Injury, poisoning and procedural complications) | 5 | 1
Traumatic haemothorax (Injury, poisoning and procedural complications) | 0 | 1
Urinary retention postoperative (Injury, poisoning and procedural complications) | 0 | 1
Wrist fracture (Injury, poisoning and procedural complications) | 0 | 1
Electrophoresis protein abnormal (Investigations) | 1 | 0
Foetal heart rate abnormal (Investigations) | 0 | 1
International normalised ratio increased (Investigations) | 1 | 0
Dehydration (Metabolism and nutrition disorders) | 1 | 3
Diabetes mellitus inadequate control (Metabolism and nutrition disorders) | 2 | 1
Diabetic ketoacidosis (Metabolism and nutrition disorders) | 5 | 1
Dyslipidaemia (Metabolism and nutrition disorders) | 1 | 0
Hypoglycaemia (Metabolism and nutrition disorders) | 1 | 0
Hypokalaemia (Metabolism and nutrition disorders) | 2 | 2
Hyponatraemia (Metabolism and nutrition disorders) | 2 | 0
Type 2 diabetes mellitus (Metabolism and nutrition disorders) | 1 | 1
Back pain (Musculoskeletal and connective tissue disorders) | 1 | 1
Bursitis (Musculoskeletal and connective tissue disorders) | 1 | 0
Costochondritis (Musculoskeletal and connective tissue disorders) | 0 | 1
Flank pain (Musculoskeletal and connective tissue disorders) | 0 | 1
Intervertebral disc degeneration (Musculoskeletal and connective tissue disorders) | 1 | 1
Intervertebral disc protrusion (Musculoskeletal and connective tissue disorders) | 1 | 0
Lumbar spinal stenosis (Musculoskeletal and connective tissue disorders) | 2 | 0
Muscular weakness (Musculoskeletal and connective tissue disorders) | 1 | 0
Musculoskeletal chest pain (Musculoskeletal and connective tissue disorders) | 1 | 0
Myositis (Musculoskeletal and connective tissue disorders) | 0 | 1
Neck pain (Musculoskeletal and connective tissue disorders) | 0 | 1
Osteoarthritis (Musculoskeletal and connective tissue disorders) | 7 | 3
Rhabdomyolysis (Musculoskeletal and connective tissue disorders) | 2 | 0
Rotator cuff syndrome (Musculoskeletal and connective tissue disorders) | 0 | 1
Spinal column stenosis (Musculoskeletal and connective tissue disorders) | 1 | 0
Spinal osteoarthritis (Musculoskeletal and connective tissue disorders) | 2 | 0
Spondylolisthesis (Musculoskeletal and connective tissue disorders) | 1 | 0
Vertebral foraminal stenosis (Musculoskeletal and connective tissue disorders) | 1 | 0
Adenocarcinoma of colon (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 | 1
Brain neoplasm benign (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 | 0
Breast cancer (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 2 | 0
Cervix carcinoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 1
Cholangiocarcinoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 1
Clear cell renal cell carcinoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 | 0
Colon adenoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 2 | 0
Ductal adenocarcinoma of pancreas (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 | 0
Endometrial cancer (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 | 0
Hodgkin's disease (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 | 0
Intraductal papillary mucinous neoplasm (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 | 0
Intraductal proliferative breast lesion (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 2 | 0
Invasive ductal breast carcinoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 2 | 0
Lung adenocarcinoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 | 0
Lung cancer metastatic (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 | 0
Malignant melanoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 | 0
Metastatic renal cell carcinoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 | 0
Oesophageal adenocarcinoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 1
Ovarian cancer stage iii (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 1
Ovarian germ cell teratoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 1
Pancreatic carcinoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 | 0
Pancreatic carcinoma metastatic (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 | 1
Papillary thyroid cancer (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 1
Pelvic neoplasm (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 | 0
Plasma cell myeloma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 | 0
Prostate cancer (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 3 | 4
Prostate cancer stage ii (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 | 0
Rectal adenocarcinoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 | 0
Small cell lung cancer metastatic (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 | 0
Squamous cell carcinoma of the cervix (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 | 0
Squamous cell carcinoma of the oral cavity (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 | 0
Uterine leiomyoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 | 2
Carotid artery stenosis (Nervous system disorders) | 2 | 1
Carotid sinus syndrome (Nervous system disorders) | 0 | 1
Cauda equina syndrome (Nervous system disorders) | 1 | 0
Cerebrovascular accident (Nervous system disorders) | 7 | 3
Cervical myelopathy (Nervous system disorders) | 1 | 1
Complex partial seizures (Nervous system disorders) | 1 | 1
Convulsion (Nervous system disorders) | 4 | 1
Dizziness (Nervous system disorders) | 2 | 0
Embolic stroke (Nervous system disorders) | 1 | 0
Haemorrhagic stroke (Nervous system disorders) | 0 | 1
Headache (Nervous system disorders) | 1 | 0
Hepatic encephalopathy (Nervous system disorders) | 1 | 0
Hypoaesthesia (Nervous system disorders) | 0 | 1
Hypoxic-ischaemic encephalopathy (Nervous system disorders) | 2 | 0
Ischaemic stroke (Nervous system disorders) | 2 | 1
Lacunar infarction (Nervous system disorders) | 1 | 0
Lumbar radiculopathy (Nervous system disorders) | 1 | 0
Migraine (Nervous system disorders) | 1 | 0
Neuropathy peripheral (Nervous system disorders) | 1 | 0
Radial nerve palsy (Nervous system disorders) | 1 | 0
Spondylitic myelopathy (Nervous system disorders) | 0 | 1
Subarachnoid haemorrhage (Nervous system disorders) | 1 | 0
Syncope (Nervous system disorders) | 2 | 4
Thalamic infarction (Nervous system disorders) | 1 | 0
Thrombotic stroke (Nervous system disorders) | 0 | 1
Transient global amnesia (Nervous system disorders) | 1 | 0
Transient ischaemic attack (Nervous system disorders) | 4 | 1
Abortion spontaneous (Pregnancy, puerperium and perinatal conditions) | 3 | 2
Foetal growth restriction (Pregnancy, puerperium and perinatal conditions) | 1 | 0
Gestational diabetes (Pregnancy, puerperium and perinatal conditions) | 1 | 0
Oligohydramnios (Pregnancy, puerperium and perinatal conditions) | 0 | 1
Placenta praevia (Pregnancy, puerperium and perinatal conditions) | 1 | 0
Bipolar disorder (Psychiatric disorders) | 3 | 1
Bipolar i disorder (Psychiatric disorders) | 4 | 0
Confusional state (Psychiatric disorders) | 0 | 1
Delirium (Psychiatric disorders) | 1 | 0
Depression (Psychiatric disorders) | 5 | 1
Depression suicidal (Psychiatric disorders) | 1 | 0
Mental status changes (Psychiatric disorders) | 3 | 1
Schizoaffective disorder (Psychiatric disorders) | 1 | 0
Schizophrenia (Psychiatric disorders) | 1 | 0
Substance-induced psychotic disorder (Psychiatric disorders) | 0 | 1
Suicidal ideation (Psychiatric disorders) | 3 | 1
Suicide attempt (Psychiatric disorders) | 3 | 1
Acute prerenal failure (Renal and urinary disorders) | 1 | 0
Bladder disorder (Renal and urinary disorders) | 0 | 1
Calculus ureteric (Renal and urinary disorders) | 4 | 2
Nephrolithiasis (Renal and urinary disorders) | 0 | 1
Prerenal failure (Renal and urinary disorders) | 1 | 0
Renal failure (Renal and urinary disorders) | 0 | 1
Renal failure acute (Renal and urinary disorders) | 4 | 3
Renal failure chronic (Renal and urinary disorders) | 2 | 0
Tubulointerstitial nephritis (Renal and urinary disorders) | 1 | 0
Urinary retention (Renal and urinary disorders) | 0 | 2
Adenomyosis (Reproductive system and breast disorders) | 0 | 2
Cystocele (Reproductive system and breast disorders) | 1 | 0
Dysfunctional uterine bleeding (Reproductive system and breast disorders) | 1 | 0
Postmenopausal haemorrhage (Reproductive system and breast disorders) | 0 | 1
Prostatitis (Reproductive system and breast disorders) | 0 | 1
Vaginal haemorrhage (Reproductive system and breast disorders) | 0 | 1
Acute respiratory distress syndrome (Respiratory, thoracic and mediastinal disorders) | 1 | 1
Acute respiratory failure (Respiratory, thoracic and mediastinal disorders) | 6 | 1
Asthma (Respiratory, thoracic and mediastinal disorders) | 5 | 1
Chronic obstructive pulmonary disease (Respiratory, thoracic and mediastinal disorders) | 9 | 3
Diaphragmatic paralysis (Respiratory, thoracic and mediastinal disorders) | 1 | 0
Diaphragmatic rupture (Respiratory, thoracic and mediastinal disorders) | 1 | 0
Dyspnoea (Respiratory, thoracic and mediastinal disorders) | 2 | 0
Haemothorax (Respiratory, thoracic and mediastinal disorders) | 1 | 0
Hiccups (Respiratory, thoracic and mediastinal disorders) | 1 | 0
Hypoxia (Respiratory, thoracic and mediastinal disorders) | 2 | 0
Lung infiltration (Respiratory, thoracic and mediastinal disorders) | 1 | 0
Nasal polyps (Respiratory, thoracic and mediastinal disorders) | 1 | 0
Pleural effusion (Respiratory, thoracic and mediastinal disorders) | 2 | 0
Pleuritic pain (Respiratory, thoracic and mediastinal disorders) | 1 | 0
Pneumonia aspiration (Respiratory, thoracic and mediastinal disorders) | 1 | 1
Pneumothorax (Respiratory, thoracic and mediastinal disorders) | 4 | 1
Pulmonary embolism (Respiratory, thoracic and mediastinal disorders) | 3 | 2
Pulmonary oedema (Respiratory, thoracic and mediastinal disorders) | 1 | 0
Respiratory arrest (Respiratory, thoracic and mediastinal disorders) | 0 | 1
Respiratory failure (Respiratory, thoracic and mediastinal disorders) | 1 | 2
Diabetic foot (Skin and subcutaneous tissue disorders) | 1 | 2
Hidradenitis (Skin and subcutaneous tissue disorders) | 1 | 0
Victim of homicide (Social circumstances) | 1 | 0
Aortic aneurysm (Vascular disorders) | 2 | 0
Aortic stenosis (Vascular disorders) | 0 | 1
Deep vein thrombosis (Vascular disorders) | 4 | 3
Hypertension (Vascular disorders) | 5 | 3
Hypertensive crisis (Vascular disorders) | 2 | 0
Hypotension (Vascular disorders) | 2 | 2
Peripheral vascular disorder (Vascular disorders) | 1 | 0
Thrombophlebitis superficial (Vascular disorders) | 1 | 0
OTHER ADVERSE EVENTS (reported when occurring in more than 1% of participants in an arm); cells are participants affected of the arm's N at risk:
Term (organ system) | HEPLISAV (N=5587) | Engerix-B (N=2781)
Acute sinusitis (Infections and infestations) | 59 | 37
Bronchitis (Infections and infestations) | 174 | 102
Sinusitis (Infections and infestations) | 149 | 84
Upper respiratory tract infection (Infections and infestations) | 191 | 92
Urinary tract infection (Infections and infestations) | 132 | 63
Type 2 diabetes mellitus (Metabolism and nutrition disorders) | 66 | 36
Arthralgia (Musculoskeletal and connective tissue disorders) | 98 | 54
Back pain (Musculoskeletal and connective tissue disorders) | 115 | 54
Musculoskeletal pain (Musculoskeletal and connective tissue disorders) | 45 | 30
Osteoarthritis (Musculoskeletal and connective tissue disorders) | 72 | 30
Pain in extremity (Musculoskeletal and connective tissue disorders) | 72 | 28
Cough (Respiratory, thoracic and mediastinal disorders) | 62 | 37
Hypertension (Vascular disorders) | 128 | 57

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
Principal Investigator may communicate study results with prior written consent from Dynavax.